CLINICAL TRIAL: NCT01482689
Title: Bioavailability of Vitamin D in Cod Liver Oil and Multivitamin Tablets in Healthy Subjects in Norway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Norwegian Institute of Public Health (Other Government); Hormone Laboratory, Aker University Hospital, Oslo, Norway (Other); Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Principal Investigator, Haakon E. Meyer, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: S-04340
Record Dates: First submitted 2011-11-23; First posted 2011-11-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Bioavailability; Vitamin D metabolism; Bone turnover
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil capsule (Experimental)
  Interventions: Dietary Supplement: Fish oil capsule (specially manufactured for the study)
- Multivitamin tablet (Experimental)
  Interventions: Dietary Supplement: Multivitamin tablet of type: Vitaplex ABCD

INTERVENTIONS:
Dietary Supplement: Fish oil capsule (specially manufactured for the study) — One capsule per day for 4 weeks (28 days). The fish oil group receives a daily supplement of one fish oil capsule, specially manufactured for the present study by Peter Möller (now Möller's, Nydalen, Norway). The fish oil capsules are aimed to contain a dose of cholecalciferol identical to the dose already found in the multivitamin tablets by analysis in an independent laboratory (AS Vitas, Oslo, Norway), and similar doses of vitamin A. In addition, the fish oil capsule contains vitamin E and n-3 fatty acids.
  Arms: Fish oil capsule
Dietary Supplement: Multivitamin tablet of type: Vitaplex ABCD — One tablet per day for 4 weeks (28 days). The multivitamin group receives a daily supplement of one multivitamin tablet of type Vitaplex ABCD (Cederroth AS, Revetal, Norway), a common vitamin supplement sold in grocery stores in Norway. In addition to 10 micrograms (400 IU) of cholecalciferol,the multivitamin tablet contains vitamin A and the water-soluble vitamins: B1, B2, B6, Niacin, pantothenic acid, and vitamin C.
  Other Names: Vitaplex ABCD
  Arms: Multivitamin tablet

SUMMARY:
The main aim of the present study is to compare the bioavailability of vitamin D from cod liver oil and multivitamin tablets given to healthy individuals under the same conditions, as well as to study the influence of gender and ethnicity on vitamin D absorption. Healthy subjects will be randomised into two parallel groups receiving 10 micrograms (400 IU) per day of vitamin D3 from one fish oil capsule or one solid multivitamin tablet, respectively. Serum samples will be drawn at baseline and after four weeks (28 days) for the analysis of 25-hydroxyvitamin D, 1,25-dihydroxyvitamin D, parathyroid hormone, and tartrate resistant acid phosphatase in serum.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to meet at baseline and follow-up visit

Exclusion Criteria:

* Using any vitamin D containing supplements regularly (> once per week)
* Travelled to sunny countries in the previous 3 months
* Used a tanning bed in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-02; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Difference in delta serum 25-hydroxyvitamin D (nmol/l) between the two parallel intervention groups | 4 weeks (28 days) between baseline and follow-up visit

SECONDARY OUTCOMES:
Difference in delta 25-hydroxyvitamin D (nmol/l) between men and women | 4 weeks (28 days) between baseline and follow-up visit
Difference in delta 25-hydroxyvitamin D (nmol/l) between ethnic groups | 4 weeks (28 days) between baseline and follow-up visit
Correlation between change in 25-hydroxyvitamin D (nmol/l) and change in serum intact parathyroid hormone (pmol/l) | 4 weeks (28 days) between baseline and follow-up visit
Correlation between change in 25-hydroxyvitamin D (nmol/l) and change in serum 1,25-dihydroxyvitamin D (pmol/l) | 4 weeks (28 days) between baseline and follow-up visit
Correlation between change in 25-hydroxyvitamin D (nmol/l) and change in serum osteoclast-specific tartrate-resistant acid phosphatase (TRACP 5b); U/l | 4 weeks (28 days) between baseline and follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

REFERENCES:
- [Result] Holvik K, Madar AA, Meyer HE, Lofthus CM, Stene LC. A randomised comparison of increase in serum 25-hydroxyvitamin D concentration after 4 weeks of daily oral intake of 10 microg cholecalciferol from multivitamin tablets or fish oil capsules in healthy young adults. Br J Nutr. 2007 Sep;98(3):620-5. doi: 10.1017/S000711450773074X. Epub 2007 Apr 24. PMID 17456248
- [Derived] Holvik K, Madar AA, Meyer HE, Lofthus CM, Stene LC. Changes in the vitamin D endocrine system and bone turnover after oral vitamin D3 supplementation in healthy adults: results of a randomised trial. BMC Endocr Disord. 2012 Jun 13;12:7. doi: 10.1186/1472-6823-12-7. PMID 22695105